CLINICAL TRIAL: NCT03453060
Title: A Phase 1, Single Ascending Dose, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of E-WE Thrombin as an Intravenous Bolus in Healthy Adult Subjects
Brief Title: Safety and Tolerability Study of E-WE Thrombin in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aronora, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EWE-17-01
Record Dates: First submitted 2018-02-20; First posted 2018-03-05 (Actual); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- E-WE Thrombin Dose 1 (Experimental): Participants will receive a single intravenous dose of 0.5 mcg/kg E-WE Thrombin.
  Interventions: Drug: E-WE Thrombin- Dose 1
- E-WE Thrombin Dose 2 (Experimental): Participants will receive a single intravenous dose of 1.0 mcg/kg E-WE Thrombin.
  Interventions: Drug: E-WE Thrombin- Dose 2
- E-WE Thrombin Dose 3 (Experimental): Participants will receive a single intravenous dose of 2.0 mcg/kg E-WE Thrombin.
  Interventions: Drug: E-WE Thrombin- Dose 3
- E-WE Thrombin Dose 4 (Experimental): Participants will receive a single intravenous dose of 4.0 mcg/kg E-WE Thrombin.
  Interventions: Drug: E-WE Thrombin- Dose 4
- Placebo (Placebo Comparator): Participants will receive a single intravenous dose of placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: E-WE Thrombin- Dose 1 — Participants received a single intravenous dose of 0.5 mcg/kg E-WE Thrombin.
  Other Names: AB002- Dose 1
  Arms: E-WE Thrombin Dose 1
Drug: E-WE Thrombin- Dose 2 — Participants received a single intravenous dose of 1.0 mcg/kg E-WE Thrombin.
  Other Names: AB002- Dose 2
  Arms: E-WE Thrombin Dose 2
Drug: E-WE Thrombin- Dose 3 — Participants received a single intravenous dose of 2.0 mcg/kg E-WE Thrombin.
  Other Names: AB002- Dose 3
  Arms: E-WE Thrombin Dose 3
Drug: E-WE Thrombin- Dose 4 — Participants received a single intravenous dose of 4.0 mcg/kg E-WE Thrombin.
  Other Names: AB002- Dose 4
  Arms: E-WE Thrombin Dose 4
Other: Placebo — Participants received a single intravenous dose of placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacodynamics of a single iv dose of E-WE Thrombin in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male and/or female (females of non-childbearing potential only), 18 to 55 years of age, inclusive, at screening.
2. Continuous non-smoker, who has not used nicotine-containing products for at least 3 months prior to dosing, based on subject self-reporting.
3. Body mass index (BMI) ≥ 18 and < 29 (kg/m2) at screening and weight between 50 and 125 kg (inclusive) at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms, as deemed by the PI or designee.
5. A female must be of non childbearing potential and must have undergone one of the following sterilization procedures at least 6 months prior to dosing:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy. or be postmenopausal with amenorrhea for at least 1 year prior to dosing and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status.
6. A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to dosing of study drug. A male who has been vasectomized less than 4 months prior to dosing must follow the same restrictions as a non vasectomized male).
7. If male, must agree to not donate sperm from dosing until 90 days after dosing.
8. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to dosing.
5. Consumes 3 units or more of alcohol per day (e.g., 1 unit is equivalent to 240 mL of wine, 1 bottle of beer [12 oz.], or 1 shot of liquor [1 oz.]).
6. History or presence of hypersensitivity or idiosyncratic reaction to the study drug and excipients or related compounds.
7. History or presence of a disease or disorder, acquired or inherited, that is active, or could be reasonably expected to become active during the study, including but not limited to:

   * Hypersensitivity to ß-lactam / penicillin derivatives;
   * Bleeding and blood coagulation disorders, including stroke, hemophilias, thrombophilias, or heparin-induced thrombocytopenia;
   * Ischemic disorders, including stroke, heart attack, coronary artery disease;
   * Gastrointestinal disorders, including gastrointestinal bleeds, gallstones, ulcers, diseases or dysfunction of the liver and excluding appendectomy and/or cholecystectomy;
   * Genitourinary disorders, including renal disease;
   * Cardiovascular disorders, including aneurysms, vasculitis;
   * All conditions that are associated with taking medications for pain;
   * Infection of any organ or system within 30 days of dosing;
   * Malignant and cancerous neoplasms of any organ or system;
   * Psychiatric and behavioral disorders;
   * A clinically significant hematological disorder of any type;
   * Inflammation and inflammatory diseases of any organ system.
8. Females of childbearing potential.
9. Females who are pregnant or who are lactating.
10. Positive urine drug or alcohol results at screening or check in.
11. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
12. Supine blood pressure is less than 90/50 mmHg or greater than 140/90 mmHg at screening.
13. Supine heart rate is lower than 40 bpm or higher than 99 bpm at screening.
14. QTcF interval > 450 msec for males or > 460 msec for females, or history of prolonged QT syndrome at screening.
15. Estimated creatinine clearance < 90 mL/minutes at screening using the Cockcroft Gault estimation.
16. Unable to refrain from or anticipates the use of:

    * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning approximately 14 days prior to dosing and throughout the study.
    * Any oral or injectable anticoagulant (e.g., warfarin, heparin, low molecular weight heparin, etc.), coagulants (aprotinin, tranexamic acid, epsilon-aminocaproic acid, and aminomethylbenzoic acid), anti-platelet (e.g., clopidogrel), nonsteroidal anti-inflammatory drugs (NSAIDs) and/or acetylsalicylic acid (ASA) beginning approximately 10 days prior to dosing and throughout the study.
    * Any drugs known to be significant inducers of cytochrome P-450 enzymes and/or P glycoprotein, including St. John's Wort, for 28 days prior to dosing and throughout the study.

    Appropriate sources (e.g., Flockhart TableTM) will be consulted to confirm lack of pharmacokinetic/ pharmacodynamic interaction with study medication. Acetaminophen (up to 2 g per 24 hour period) or any other treatment of an adverse event, drug related or not, and considered appropriate and allowable by the PI or designee may be permitted after dosing.
17. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 30 days prior to dosing and throughout the study.
18. Has participated in strenuous exercise or physical activity within 72 hours prior to Day 1, unless deemed acceptable by the PI or designee.
19. Donation of blood or significant blood loss within 56 days prior to dosing.
20. Plasma donation within 7 days prior to dosing.
21. Has been hospitalized within 2 months of Day -1.
22. Participation in another clinical study within 30 days prior to dosing. The 30-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study.
23. Surgery within the past 90 days prior to dosing which in the opinion of the PI or designee is clinically relevant.
24. Presence of any scars, or tattoos which may obscure the injection site, as deemed by PI or designee.
25. Any condition or circumstance, in the opinion of the PI or designee, which may make the subject unlikely to complete the study or comply with study procedures and requirements, or may pose a risk to the subject's safety.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tucker EI, Verbout NG, Markway BD, Wallisch M, Lorentz CU, Hinds MT, Shatzel JJ, Pelc LA, Wood DC, McCarty OJT, Di Cera E, Gruber A. The protein C activator AB002 rapidly interrupts thrombus development in baboons. Blood. 2020 Feb 27;135(9):689-699. doi: 10.1182/blood.2019002771. PMID 31977000

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 132 participants were screened for the study, of which 111 did not meet eligibility criteria, declined to participate, or were dropped alternates. The remaining 21 participants were randomized into the study, with each dose level occurring in sequential order.
Groups:
- E-WE Thrombin Dose 1: Participants received a single intravenous dose of 0.5 mcg/kg E-WE Thrombin.
- E-WE Thrombin Dose 2: Participants received a single intravenous dose of 1.0 mcg/kg E-WE Thrombin.
- E-WE Thrombin Dose 3: Participants received a single intravenous dose of 2.0 mcg/kg E-WE Thrombin.
- E-WE Thrombin Dose 4: Participants received a single intravenous dose of 4.0 mcg/kg E-WE Thrombin.
Period: Overall Study
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Started | 4 | 4 | 4 | 4 | 5
Completed | 4 | 4 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5 | 21
Age, Continuous [Mean (Full Range); unit: years] | 44.0 [40 to 52] | 37.3 [26 to 47] | 33.8 [23 to 46] | 36.0 [23 to 52] | 43.0 [33 to 53] | 39.0 [23 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 3 | 4 | 14
  Male | 1 | 2 | 2 | 1 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 2 | 3 | 4 | 16
  Not Hispanic or Latino | 1 | 0 | 2 | 1 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 0 | 2
  White | 3 | 3 | 3 | 4 | 5 | 18
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With Treatment-emergent Adverse Events (TEAEs) Will be Summarized Using Frequency Counts.
Description: TEAEs will be determined by symptom driven physical examinations that can include assessment of the skin, head, ears, eyes, nose, throat, respiratory system, cardiovascular system, gastrointestinal system, neurological condition, blood and lymphatic systems, and the musculoskeletal system.
Time Frame: one month
Population: Subjects who received any dose of study drug or placebo were included in the as-treated population and subjects were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 3 | 1

2. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Body Temperature, Frequency, and Relation to Treatment Will be Assessed.
Description: Body temperature will be measured in degrees Celsius. Clinically significant changes in body temperature are determined by the PI or designee.
Time Frame: two days
Population: Subjects who had received any dose of study drug or placebo were included in the as-treated population and subjects were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Respiratory Rate, Frequency, and Relation to Treatment Will be Assessed.
Description: Respiratory rate will be measured in breaths per minute. Clinically significant changes in respiratory rate are determined by the PI.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Blood Pressure (Systolic and Diastolic), Frequency, and Relation to Treatment Will be Assessed.
Description: Systolic and diastolic blood pressure will be measured in mmHg. Clinically significant changes in systolic and diastolic blood pressure are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Heart Rate, Frequency, and Relation to Treatment Will be Assessed.
Description: Heart rate will be measured in beats per minute. Clinically significant changes in heart rate are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: The Number of Subjects With Abnormal Electrocardiogram and Frequency and/ or Adverse Events That Are Related to Treatment.
Description: 12-lead electrocardiogram measurement. Abnormal electrocardiograms are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Activated Partial Thromboplastin Time (aPTT), Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Coagulation Panel.
Description: Plasma aPTT will be measured in seconds. Clinically significant changes in aPTT are determined by the PI or designee.
Time Frame: one month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Prothrombin Time, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Coagulation Panel.
Description: Prothrombin time will be measured in seconds. Clinically significant changes in prothrombin time are determined by the PI or designee.
Time Frame: one month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Thrombin Time, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Coagulation Panel.
Description: Thrombin time will be measured in seconds. Clinically significant changes in thrombin time are determined by the PI or designee.
Time Frame: one month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Plasma Fibrinogen, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Coagulation Panel.
Description: Plasma fibrinogen levels will be measured in mg/dL. Clinically significant changes in plasma fibrinogen levels are determined by the PI or designee.
Time Frame: one month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: The Number of Subjects With Injection Site Reaction and/ or Adverse Events That Are Related to Treatment.
Description: Injection site reaction assessment (pain, tenderness, erythema/ redness, and induration/ swelling.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: The Number of Subjects That Develop Treatment-related Immunogenicity.
Description: Immunogenicity measured by plasma anti-drug antibodies.
Time Frame: one month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Blood Urea Nitrogen Levels (BUN) as Part of a Standard Serum Chemistry Panel, Frequency, and Relation to Treatment Will be Assessed.
Description: BUN levels in the blood will be measured in mg/dL. Clinically significant changes in BUN are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Bilirubin (Total and Direct) Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Bilirubin (total and direct) levels in the blood will be measured in mg/dL. Clinically significant changes in total and direct bilirubin levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Alkaline Phosphatase Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Alkaline phosphatase levels in the blood will be measured in U/L. Clinically significant changes in alkaline phosphatase levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Aspartate Aminotransferase (AST) Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: AST levels in the blood will be measured in U/L. Clinically significant changes in AST levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Alanine Aminotransferase (ALT) Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: ALT levels in the blood will be measured in U/L. Clinically significant changes in ALT levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Lactate Dehydrogenase (LDH) Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: LDH levels in the blood will be measured in U/L. Clinically significant changes in LDH levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Albumin Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Albumin levels in the blood will be measured in g/dL. Clinically significant changes in albumin levels are determined by the PI or designee.
Time Frame: two days.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

20. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Sodium Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Sodium levels will be measured in mEq/L. Clinically significant changes in sodium levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

21. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Potassium Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Potassium levels will be measured in mEq/L. Clinically significant changes in potassium levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

22. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Chloride Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Chloride levels will be measured in mEq/L. Clinically significant changes in chloride levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

23. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Bicarbonate Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Bicarbonate levels will be measured in mEq/L. Clinically significant changes in bicarbonate levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

24. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Glucose Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Blood glucose levels will be measured in mg/dL. Clinically significant changes in blood glucose levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

25. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Creatinine Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Creatinine levels will be measured in mg/dL. Clinically significant changes in creatinine levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

26. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Hemoglobin Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Hemoglobin levels will be measured in g/dL. Clinically significant changes in hemoglobin levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

27. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Hematocrit Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Hematocrit levels will be measured in %. Clinically significant changes in hematocrit levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

28. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Total Leukocyte Counts, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Total leukocyte counts will be measured in 10˄3/uL. Clinically significant changes in leukocyte counts are determined by the PI or designee.
Time Frame: two days.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

29. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Differential Leukocyte Counts, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Differential leukocyte counts will be measured in %. Clinically significant changes in differential leukocyte counts are determined by the PI or designee.
Time Frame: two days.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

30. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Red Blood Cell Count, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Red blood cell count will be measured in 10˄6/uL. Clinically significant changes in red blood cell counts are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

31. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Platelet Count, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Platelet count will be measured in 10˄3/uL. Clinically significant changes in platelet counts are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

32. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine pH, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel.
Description: pH of the urine will be measured. Clinically significant changes in urine pH are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

33. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Specific Gravity, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel.
Description: Specific gravity of the urine will be evaluated. Clinically significant changes in specific gravity are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

34. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Protein Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel.
Description: Protein levels in the urine will be evaluated. Clinically significant changes in protein levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

35. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Glucose Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel.
Description: Glucose levels in the urine will be evaluated. Clinically significant changes in urine glucose are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

36. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Ketone Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel.
Description: Ketone levels in the urine will be evaluated. Clinically significant changes in urine ketone levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

37. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Bilirubin Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel.
Description: Bilirubin levels in the urine will be evaluated. Clinically significant changes in urine bilirubin levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

38. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Blood Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel.
Description: Blood levels in the urine will be evaluated. Clinically significant changes in urine blood levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

39. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Nitrite Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel.
Description: Nitrite levels in the urine will be evaluated. Clinically significant changes in urine nitrite levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

40. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Urobilinogen Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel.
Description: Urobilinogen levels in the urine will be evaluated. Clinically significant changes in urine urobilinogen levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

41. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Leukocyte Esterase Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel.
Description: Leukocyte esterase levels in the urine will be evaluated. Clinically significant changes in urine leukocyte esterase levels are determined by the PI or designee.
Time Frame: two days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

42. Secondary Outcome: The Effect of a Single Intravenous Dose of E-WE Thrombin on Generation of Activated Protein C- Protein C Inhibitor Complexes (APC-PCI).
Description: Plasma APC-PCI levels will be measured in ng/mL.
Time Frame: Predose, 0.08, 0.25, 0.5, 1, 2, 4, and 24h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
ng/mL
  predose | 1.8 (0.9) | 1.3 (0.7) | 2.0 (0.7) | 1.0 (0.0) | 1.5 (0.7)
  0.08 hours post dose | 61.8 (16.3) | 123.0 (5.0) | 195.3 (16.8) | 283.3 (61.2) | 1.7 (0.9)
  0.25 hours post dose | 108.2 (20.5) | 218.3 (4.6) | 364.8 (86.4) | 579.0 (82.0) | 1.2 (0.5)
  0.5 hours post dose | 122.0 (18.6) | 229.8 (19.4) | 470.8 (140.9) | 678.3 (84.8) | 1.3 (0.6)
  1 hour post dose | 90.9 (12.9) | 194.5 (24.2) | 328.8 (94.0) | 480.5 (33.6) | 1.2 (0.5)
  2 hours post dose | 27.3 (3.8) | 56.2 (14.8) | 124.5 (40.4) | 132.3 (17.4) | 1.2 (0.5)
  4 hours post dose | 3.5 (0.5) | 5.9 (1.3) | 12.7 (6.2) | 15.2 (4.3) | 1.0 (0.0)
  24 hours post dose | 1.0 (0.0) | 1.0 (0.0) | 1.7 (0.9) | 1.0 (0.0) | 1.6 (0.8)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from subject check-in through follow up which occurred on Day 28.
Description: Subjects were monitored throughout confinement for adverse reactions to the study drug and/or procedures. Subjects were asked how they are feeling and were encouraged to report AEs during confinement and at each follow-up visit.
Arm/Group | E-WE Thrombin Dose 1 | E-WE Thrombin Dose 2 | E-WE Thrombin Dose 3 | E-WE Thrombin Dose 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 3/4 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-WE Thrombin Dose 1 (N=4) | E-WE Thrombin Dose 2 (N=4) | E-WE Thrombin Dose 3 (N=4) | E-WE Thrombin Dose 4 (N=4) | Placebo (N=5)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Aronora, Inc. shall retain title to and the right to publish all documentation, records, raw data, specimens, or other work product generated in connection with this study. Such publications shall not be made by the PI or Celerion without the prior written consent of Aronora, Inc.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT03453060/SAP_000.pdf
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT03453060/Prot_001.pdf